CLINICAL TRIAL: NCT00414609
Title: A 36-week, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Including a 2 Year Extension Study to Evaluate Efficacy and Safety of Aliskiren on the Prevention of Left Ventricular Remodeling in High Risk Post-acute Myocardial Infarction Patients When Added to Optimized Standard Therapy
Brief Title: Safety and Efficacy of Aliskiren in Post Myocardial Infarction Patients (ASPIRE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2340; NCT00699075 (obsolete NCT alias)
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction, aliskiren, heart failure; Post acute myocardial infarction with systolic dysfunction
MeSH Terms: conditions — Myocardial Infarction; Heart Failure | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren (Experimental): Core Study: Aliskiren ascending doses: 75 mg tablet for 1st week, 150 mg for 2nd week, 300 mg for next 34 weeks orally once daily in the morning.
  Extension Study: Patients from both the core arms who completed core study and signed informed consent form were included in this arm of extension study.
  Patients received 150 mg aliskiren tablet orally once a day for two weeks. Patients were then up-titrated to 300 mg aliskiren orally once a day at the discretion of the principal investigator based on their clinical condition for the duration of the study.
  Interventions: Drug: Aliskiren
- placebo (Placebo Comparator): Core study: placebo for 36 weeks once daily in the morning
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aliskiren — Aliskiren was available in 75 mg tablet, 150 mg tablet
  Other Names: Tekturna®
  Arms: Aliskiren
Drug: placebo — Placebo tablets matching aliskiren for 36 weeks once daily in the morning for core period only.
  Arms: placebo

SUMMARY:
The core and extension studies assessed the safety and efficacy of aliskiren when added to optimized standard therapy in patients that have had a high risk acute myocardial infarction (heart attack).

ELIGIBILITY:
Core Study Inclusion Criteria:

* Male or female patients 18 years and older.
* Patients within 7-42 days of an acute myocardial infarction associated with left ventricular systolic dysfunction.
* Documented left ventricular systolic dysfunction associated with the qualifying acute myocardial.
* Patients must be on stable doses of the following concomitant medications for at least 2 weeks prior to Visit 1 unless contraindicated due to intolerance:

  * A Beta-blocker
  * An Anti-platelet agent
  * A Statin
  * An evidence-based dose of an Angiotensin Converting Enzyme Inhibitor (ACEI) or Angiotensin Receptor Blocker (ARB) but not both.
* Qualifying Echocardiogram at Visit 1:

Core Study Exclusion Criteria:

* Patients requiring both Angiotensin Converting Enzyme Inhibitor (ACEI) and Angiotensin Receptor Blocker (ARB) combination therapy at V1 or any time during the study.
* Severe refractory hypertension defined as mean sitting systolic blood pressure (MSSBP) ≥ 180 mmHg and/or mean sitting diastolic blood pressure (MSDBP) ≥ 110 mmHg) at Visit 2.
* Cardiogenic shock or systolic BP < 100 mmHg or diastolic < 60 mmHg within the 24 hours prior to Visits 1 or 2
* Estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1.73m2 using the MDRD formula at Visit 1.
* Stroke or transient ischemic event (TIA) within 6 months of Study Visit 1

Extension Study Inclusion Criteria:

* Male or female patients who completed the core study through Visit 10 while on double-blind study drug
* Patients who were able to participate in the study, and who consented to do so after the purpose and nature of the study had been clearly explained to them (written informed consent)

Extension Study Exclusion Criteria:

* New York Heart Association (NYHA) class IV Congestive Heart Failure at Visit 1 (Core study Visit 10)
* Symptomatic hypotension or reported systolic blood pressure (BP) < 90 mmHg within 24 hours prior to Visit 1 (Core study Visit 10)
* Known Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73m^2 using the Modification of Diet in Renal Disease (MDRD) formula at Visit 1 (Core study Visit 10)
* Pregnant or nursing (lactating) women, where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant Unless post-menopausal or using an acceptable method of contraception
* Any surgical or medical condition that in the opinion of the investigator may place the patient at higher risk from his/her participation in the study or was likely to prevent the patient from complying with the requirements or completing the study

Other protocol-defined inclusion/exclusion criteria applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis US, Study Chair — Novartis
Locations (23):
- Novartis US, Novartis US, New Jersey, United States
- Novartis Argentina, Novartis Argentina, Argentina
- Novartis Belgium, Novartis Belgium, Belgium
- Novartis Canada, Novartis Canada, Canada
- Novartis de Colombia S.A., Bogotá, Colombia
- Novartis Czech Republic, Prague, Praha 3, Czechia
- Novartis Denmark, Novartis Denmark, Denmark
- Novartis Germany, Novartis Germany, Germany
- Novartis Hungary, Budapest, Budapest, Hungary
- Novartis Healthcare Private Limited, Worli, Mumbai, India
- Novartis Pharma, Petah Tikva, Petach Tikva, Israel
- Novartis Italy, Novartis Italy, Italy
- Novartis Netherlands, Novartis Netherlands, Netherlands
- Novartis Norway, Novartis Norway, Norway
- Novartis Poland Sp. z o.o., Warsaw, Poland
- Novartis Russia, Novartis Russia, Russia
- Novartis Slovakia, Bratislava, Bratislava Region, Slovakia
- Novartis Korea Ltd., Seoul, Seoul, South Korea
- Novartis Spain, Novartis Spain, Spain
- Novartis Sweden, Novartis Sweden, Sweden
- Novartis Turkey, Istanbul, Istanbul, Turkey (Türkiye)
- Novartis UK, Novartis, United Kingdom
- Novartis de Venezuela, S.A., Caracas, Venezuela

REFERENCES:
- [Derived] Solomon SD, Shin SH, Shah A, Skali H, Desai A, Kober L, Maggioni AP, Rouleau JL, Kelly RY, Hester A, McMurray JJ, Pfeffer MA; Aliskiren Study in Post-MI Patients to Reduce Remodeling (ASPIRE) Investigators. Effect of the direct renin inhibitor aliskiren on left ventricular remodelling following myocardial infarction with systolic dysfunction. Eur Heart J. 2011 May;32(10):1227-34. doi: 10.1093/eurheartj/ehq522. Epub 2011 Feb 10. PMID 21317148

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo_Core: Placebo for 36 weeks once daily in the morning
- Aliskiren_Core: Aliskiren ascending doses: 75 mg tablet for 1st week, 150 mg for 2nd week, 300 mg for the next 34 weeks orally once daily in the morning.
- Aliskiren_Extension: Patients from both the arms of the core study who completed core study and signed informed consent form were included in this arm of extension study.
  Patients received 150 mg aliskiren tablet orally once a day for two weeks. Patients were then up-titrated to 300 mg aliskiren orally once a day at the discretion of the principal investigator based on their clinical condition for the duration of the study.
Period: Core Study
Arm/Group | Placebo_Core | Aliskiren_Core | Aliskiren_Extension
Started | 397 | 423 | 0
Received Study Drug | 397 | 422 | 0
Echocardiogram Evaluable Set | 330 | 343 | 0
Completed | 363 | 378 | 0
Not Completed | 34 | 45 | 0
Not completed — Adverse Event | 9 | 11 | 0
Not completed — Abnormal laboratory values | 0 | 1 | 0
Not completed — Abnormal test procedure results | 1 | 1 | 0
Not completed — Protocol deviation | 0 | 1 | 0
Not completed — Patient withdrew consent | 10 | 11 | 0
Not completed — Lost to Follow-up | 7 | 4 | 0
Not completed — Administrative problems | 0 | 2 | 0
Not completed — Death | 7 | 14 | 0
Period: Extension Study
Arm/Group | Placebo_Core | Aliskiren_Core | Aliskiren_Extension
Started | 0 | 0 | 422 (Patients of both core arms who completed core study and signed informed consent form for extension.)
Echocardiogram (ECHO) Analysis Set | 0 | 0 | 400
Completed | 0 | 0 | 365
Not Completed | 0 | 0 | 57
Not completed — Adverse Event | 0 | 0 | 14
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 13
Not completed — Lost to Follow-up | 0 | 0 | 10
Not completed — Administrative problems | 0 | 0 | 1
Not completed — Death | 0 | 0 | 17

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo for 36 weeks once daily in the morning
- Aliskiren: Aliskiren ascending doses: 75 mg tablet for 1st week, 150 mg for 2nd week, 300 mg for the next 34 weeks orally once daily in the morning.
- Total: Total of all reporting groups
Arm/Group | Placebo | Aliskiren | Total
Number analyzed (Participants) | 397 | 423 | 820
Age Continuous [Mean (Standard Deviation); unit: years] — Demographics were measured for core randomized population
  years | 59.4 (11.67) | 60.7 (11.63) | 60.0 (11.66)
Age, Customized [Number; unit: Participants]
  < 65 years | 261 | 254 | 515
  ≥ 65 years and < 75 years | 93 | 114 | 207
  ≥ 75 years | 43 | 55 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 80 | 141
  Male | 336 | 343 | 679

OUTCOME MEASURES:

1. Primary Outcome: Core Study: Change From Baseline in Left Ventricular End Systolic Volume (LVESV) as Measured by Echocardiography at End of Study.
Description: Change from baseline to end of study in left ventricular end systolic volume (LVESV) as measured by echocardiography. LVESV is a measurement of the volume of blood in the heart's left ventricular chamber at the end of the heart's contraction. This measurement was made by the echocardiography lab. LVESV values between 22 to 58 mL for men and 19-49 mL for women are considered normal. Baseline LVESV was a covariate.
Time Frame: Baseline and final visit (after 26 to 36 weeks of treatment)
Population: Echocardiogram evaluable set (patients who had acceptable echocardiogram measurements both at baseline and at post-baseline after receiving at least 26 weeks of treatment)
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo_Core | Aliskiren_Core
Number analyzed (Participants) | 329 | 343
mL | -3.14 (1.01) | -4.13 (0.97)

2. Secondary Outcome: Core Study: Time to First Occurrence for the Composite Endpoints of Echocardiogram and Adjudicated Outcomes
Description: Composite outcome 1 included: Cardiovascular (CV) Death, hospitalization for heart failure (HF), or absolute reduction in Left Ventricular Ejection Fraction (LVEF) greater than 6%. Composite outcome 2 included: CV Death, hospitalization for HF, recurrent Myocardial Infarction, Stroke, or Resuscitated Sudden Death. LVEF was measured at baseline and final visit. All other events were adjudicated by a blinded external committee. Each composite endpoint analysis was based on (a) the percent of patients with that endpoint and (b) days in study to 1st event (or last exposure if no event occurred).
Time Frame: LVEF was measured at baseline and at final visit (after 26 to 36 weeks of treatment). Other endpoint components were assessed from randomization until the end of the study (week 36).
Population: Full Analysis Set (FAS) - All randomized patients who either (a) received study drug or (b) did not receive study drug but were not disqualified from randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo_Core | Aliskiren_Core
Number analyzed (Participants) | 397 | 423
Percentage of participants
  Composite Outcome 1 | 6.0 | 6.9
  Composite Outcome 2 | 8.6 | 9.2

3. Secondary Outcome: Core Study: Change From Baseline in Left Ventricular End Diastolic Volume (LVEDV)
Description: Change from baseline to end of study in left ventricular end diastolic volume (LVEDV) as measured by echocardiography. (LVEDV) is a measurement of the volume of blood in the heart's left ventricular chamber at the beginning of the chamber's filling with blood. This measurement was made by the echocardiography lab. LVEDV values between 67 to 155 mL for men and 56 to 104 mL for women are considered normal. Baseline LVEDV was a covariate.
Time Frame: Baseline and final visit (after 26 to 36 weeks of treatment)
Population: Echocardiogram evaluable set: Patients who had acceptable echocardiogram measurements both at baseline and at post-baseline after receiving at least 26 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo_Core | Aliskiren_Core
Number analyzed (Participants) | 329 | 343
mL | -1.37 (1.19) | -3.08 (1.15)

4. Secondary Outcome: Core Study: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: Change from baseline to end of study in left ventricular ejection fraction (LVEF) (%) as measured by echocardiography. LVEF is the fraction of blood (in percent) pumped out of the heart's left ventricular chamber with each heart beat, and is a measure of cardiac output for the heart. This measurement was made by the echocardiography lab. Ejection fraction percentages > 55% are considered normal. Baseline LVEF was a covariate.
Time Frame: Baseline and final visit (after 26 to 36 weeks of treatment )
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent of blood pumped from LV chamber
Arm/Group | Placebo_Core | Aliskiren_Core
Number analyzed (Participants) | 329 | 343
percent of blood pumped from LV chamber | 2.12 (0.27) | 2.24 (0.26)

5. Secondary Outcome: Core Study: Change From Baseline to End of Study in Infarction Segment Length (ISL) as Measured by Echocardiography
Description: Change from baseline to end of study in infarction segment length (ISL) (%) as measured by echocardiography. This is the length of the myocardial infarction segment as a percentage of the total cavity perimeter length as calculated by the echocardiography lab. Baseline ISL was a covariate.
Time Frame: Baseline and final visit (after 26 to 36 weeks of treatment)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent of total cavity perimeter length
Arm/Group | Placebo_Core | Aliskiren_Core
Number analyzed (Participants) | 330 | 343
percent of total cavity perimeter length | -4.30 (0.53) | -5.04 (0.51)

6. Secondary Outcome: Core Study: Change From Baseline to End of Study in Wall Motion Score (WMS) as Measured by Echocardiography
Description: Change from baseline to end of study in Wall Motion Score (WMS) as measured by echocardiography. WMS was obtained by examining multiple segments of the left ventricle and assigning each segment a score based on myocardial thickening: 1 for normal, 2 for hypokinetic; 3 for akinetic; and 4 for dyskinetic. The WMS was obtained as the average score for the segments visualized and was calculated by the echocardiography lab. Possible values range from 1 to 5. Higher scores are considered worse. Baseline WMS was a covariate.
Time Frame: Baseline and final visit (after 26 to 36 weeks of treatment)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo_Core | Aliskiren_Core
Number analyzed (Participants) | 327 | 340
Scores on a scale | -0.08 (0.01) | -0.10 (0.01)

7. Primary Outcome: Extension Study: Percentage of Participants With Deaths, Serious Adverse Events (SAEs), Discontinuation for Adverse Events (AEs) and Discontinuations for Abnormal Lab Values
Description: AEs are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: Extension study (24 weeks)
Population: Extension Population (considered as Safety population) consisting of all enrolled patients who received at least one dose of study medication in the extension study.
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren_Extension
Number analyzed (Participants) | 422
Percentage of participants
  Deaths | 4.0
  SAEs | 29.9
  AE discontinuations | 7.1
  Drug-related AE discontinuations | 2.4
  SAE discontinuations | 5.2
  Discontinuations for abnormal lab values | 0

8. Secondary Outcome: Extension Study: Change From Baseline in Left Ventricular End Systolic Volume (LVESV) at Month 12
Description: Change from baseline to Month 12 in left ventricular end systolic volume (LVESV) as measured by echocardiography. LVESV is a measurement of the volume of blood in the heart's left ventricular chamber at the end of the heart's contraction. This measurement was made by the echocardiography lab. LVESV values between 22 to 58 mL for men and 19-49 mL for women are considered normal.
Time Frame: Baseline(extension study), Month 12 (extension study)
Population: Echocardiogram Analysis Set consisting of all patients in the extension population who had acceptable ECHO measurements at extension baseline and Month 12.
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Aliskiren_Extension
Number analyzed (Participants) | 302
Milliliter (mL) | -6.2 (14.32)

9. Secondary Outcome: Extension Study: Change From Baseline in Left Ventricular End Diastolic Volume (LVEDV) at Month 12
Description: Change from baseline to Month 12 in left ventricular end diastolic volume (LVEDV) as measured by echocardiography. LVEDV is a measurement of the volume of blood in the heart's left ventricular chamber at the beginning of the chamber's filling with blood. This measurement was made by the echocardiography lab. LVEDV values between 67 to 155 mL for men and 56 to 104 mL for women are considered normal.
Time Frame: Baseline (extension study), Month 12 (extension study)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Groups:
- Aliskiren_Extension: 150 mg aliskiren tablet orally once a day for two weeks. Patients were then up-titrated to 300 mg aliskiren orally once a day at the discretion of the principal investigator based on their clinical condition for the duration of the study.
Arm/Group | Aliskiren_Extension
Number analyzed (Participants) | 302
Milliliter (mL) | 6.0 (18.34)

10. Secondary Outcome: Extension Study: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Month 12
Description: Change from baseline to Month 12 in left ventricular ejection fraction (LVEF) (%) as measured by echocardiography. LVEF is the fraction of blood (in percent) pumped out of the heart's left ventricular chamber with each heart beat, and is a measure of cardiac output for the heart. This measurement was made by the echocardiography lab. Ejection fraction percentages > 55% are considered normal.
Time Frame: Baseline(extension study), Month 12 (extension study)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent of blood pumped from LV chamber
Arm/Group | Aliskiren_Extension
Number analyzed (Participants) | 302
percent of blood pumped from LV chamber | 7.4 (6.46)

11. Secondary Outcome: Extension Study: Percentage of Participants With Orthostatic Blood Pressure Change
Description: Orthostatic blood pressure change is defined as a decrease of at least 20 mmHg in systolic blood pressure or a decrease of at least 10 mmHg in diastolic blood pressure when a patient moves from a sitting position to a standing position. A patient could show orthostatic blood pressure change at more than one visit. End of study is Month 24 or early discontinuation.
Time Frame: Baseline (Day 0 Extension study), Week 2, Months 1, 3, 6, 9,16, 20, 24
Population: Extension population (considered as Safety population) consisted of all enrolled patients who received at least one dose of study medication in the extension study. "n" in each of the categories is the number of participants with data available at the given time-point.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren_Extension
Number analyzed (Participants) | 422
Percentage of Participants
  Baseline (n=420) | 2.4
  Week 2 (n=416) | 4.6
  Month 1 (n=418) | 4.1
  Month 3 (n=410) | 4.6
  Month 6 (n=400) | 3.3
  Month 9 (n=397) | 4.3
  Month 12 (n=385) | 3.6
  Month 16 (n=383) | 5.0
  Month 20 (n=350) | 4.3
  Month 24 (n=360) | 3.6
  End of Study (n=422) | 3.8
  Any post-baseline visit (n=422) | 23.5

12. Secondary Outcome: Extension Study: Percentage of Participants With Specified Criteria in Selected Labs by Laboratory Parameter
Description: Fasting blood samples were collected throughout the study and were analyzed at a central laboratory. Percentage of participants with the following clinically significant laboratory values are reported:
  Potassium <3.5 mmol/L; Low value (Normal reference range: 3.5- 5.3)
  Potassium >5.5 mmol/L and Potassium >6.0 mmol/L; High values (Normal reference range: 3.5-5.3)
  Creatinine >176.8 μmol/L; High value (Normal reference range= Male: 62- 106 and Female 44- 80)
  Blood Urea Nitrogen (BUN) >14.28; High value (Normal reference range: 2.1- 8.9)
Time Frame: 24 Months
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren_Extension
Number analyzed (Participants) | 422
Percentage of participants
  Potassium <3.5 mmol/L (n=409) | 1.5
  Potassium >5.5 mmol/L (n=409) | 11.2
  Potassium ≥6.0 mmol/L (n=409) | 4.6
  Creatinine >176.8 μmol/L (n=412) | 4.4
  BUN >14.28 mmol/L (n=412) | 8.7

ADVERSE EVENTS:
Description: Core Safety population: All patients that received at least one dose of study drug.
  Extension Safety Population: All enrolled patients who received at least one dose of study medication in the extension study.
  Extension study enrolled patients from both the arms of core who complete core study and signed an informed consent form.
Arm/Group | Placebo_core | Aliskiren_core | Aliskiren_extension
Serious Adverse Events (participants affected / at risk) | 92/397 | 107/422 | 126/422
Other Adverse Events (participants affected / at risk) | 118/397 | 161/422 | 123/422
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo_core (N=397) | Aliskiren_core (N=422) | Aliskiren_extension (N=422)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 3 | 3
Acute myocardial infarction (Cardiac disorders) | 4 | 6 | 6
Angina pectoris (Cardiac disorders) | 15 | 13 | 15
Angina unstable (Cardiac disorders) | 8 | 9 | 4
Arrhythmia (Cardiac disorders) | 2 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 3
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 2 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2 | 2
Cardiac failure (Cardiac disorders) | 14 | 18 | 9
Cardiac failure acute (Cardiac disorders) | 2 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 5
Cardiac failure congestive (Cardiac disorders) | 4 | 3 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0 | 2
Coronary artery insufficiency (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 4 | 1 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 5 | 7 | 6
Myocardial ischaemia (Cardiac disorders) | 2 | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Apparent death (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 1
Death (General disorders) | 0 | 1 | 0
Device failure (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 6 | 7 | 7
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 2 | 0
Sudden death (General disorders) | 1 | 2 | 4
Thrombosis in device (General disorders) | 0 | 0 | 2
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Peritoneal abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 5 | 7 | 3
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 2 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 2 | 2 | 2
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thrombosis in device (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 2
Blood potassium increased (Investigations) | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 1 | 0 | 0
Renal function test abnormal (Investigations) | 0 | 0 | 1
Venous pressure jugular increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carcinoid tumour of the pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Basilar artery occlusion (Nervous system disorders) | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 2
Cerebral microangiopathy (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 5 | 5
Dizziness (Nervous system disorders) | 1 | 2 | 1
Encephalomalacia (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 2 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Parkinsonism (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 2 | 2 | 6
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 2 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 2 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 1
Angiopathy (Vascular disorders) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 3 | 1 | 3
Intermittent claudication (Vascular disorders) | 1 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo_core (N=397) | Aliskiren_core (N=422) | Aliskiren_extension (N=422)
Angina pectoris (Cardiac disorders) | 23 | 24 | 19
Cardiac failure (Cardiac disorders) | 21 | 30 | 7
Non-cardiac chest pain (General disorders) | 15 | 22 | 19
Nasopharyngitis (Infections and infestations) | 24 | 23 | 28
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 22 | 12
Dizziness (Nervous system disorders) | 15 | 27 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 27 | 15
Hypotension (Vascular disorders) | 16 | 36 | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.